CLINICAL TRIAL: NCT06554145
Title: Development and Evaluation of AI Program for Predicting Bacterial Species From Urine Gram Stain Specimens
Status: Recruiting | Type: Observational
Sponsor: GramEye (Industry)
Collaborators: Keio University (Other); Kameda Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: GE003
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum and other specimen used for microbiologic testing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to develop an AI that estimates bacterial species from Gram staining images of urine specimens, and to evaluate the accuracy and labor reduction effect of Gram staining Automation system equipped with this AI.

ELIGIBILITY:
Inclusion Criteria:

* Specimens for which urine culture and urine Gram staining tests were performed for clinical purposes

Exclusion Criteria:

* Samples for which suspension of use has been requested

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Specimens that have undergone urine culture and urine Gram staining for clinical purposes will be included.
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Rate of concordance between AI-estimated results with actual culture results regarding urine Gram stain specimens | Day1
  Evaluate the concordance rate between bacterial species estimation results and culture results obtained using the automatic Gram staining device with an AI program installed for analyzing urine Gram stain specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Keio University Hospital, Shinjuku-Ku, Tokyo, Japan